CLINICAL TRIAL: NCT04017403
Title: Probiotics Oral Administration Attenuate Postoperative Cognition Decline in Elderly Orthopedic Patients
Brief Title: Probiotics Attenuate Postoperative Cognition Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PAPOCD
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Necrosis of Femoral Head; Knee Osteoarthritis; Fracture of Neck of Femur; Lumbar Disc Herniation
Keywords: postoperative cognitive dysfunction; postopeartive delirium; Probiotics
MeSH Terms: conditions — Osteoarthritis, Knee; Femoral Neck Fractures; Intervertebral Disc Displacement; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): The probiotic group was treated with Bifidobacterium tripleis,one day before surgery to the sixth day after surgerythe drug is taken orally, 4 capsules at a time, 2 times a day.
  Interventions: Drug: Bifidobacterium triple live capsule
- Placebo group (Placebo Comparator): The control group was given the same package of placebo,one day before surgery to the sixth day after surgery. The drug is taken orally, 4 capsules at a time, 2 times a day.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Bifidobacterium triple live capsule — Bifidobacterium triple live capsules, indications for acute and chronic diarrhea and constipation caused by intestinal flora imbalance, can also be used for the treatment of mild to moderate acute diarrhea, chronic diarrhea and indigestion, bloating, and adjuvant treatment of intestinal flora Endotoxemia caused by disorders.
  Other Names: Peifei Kang Capsule
  Arms: Probiotic group
Drug: Placebos — Placebos were administrated as same as the bifidobacterium live capsule
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
The aim of this study was to evaluate whether perioperative probiotics can reduce the incidence of postoperative cognitive dysfunction and postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

1. . Age is greater than or equal to 65 years old
2. . Can communicate normally
3. . Selective knee ankle, hip replacement or lumbar open reduction and internal fixation under general anesthesia
4. . ASA graded at I-II level
5. . Patient or family informed consent

Exclusion Criteria:

1. . Have a brain disease, or have a history of brain disease
2. .MMSE check of less than 24 points.
3. . History of neurological and psychological disorders including AD, stroke, psychosis
4. . Serious hearing or visual impairment
5. . Preoperative systolic blood pressure >190mmhg, or diastolic blood pressure >100mmhg
6. . The patient or family refuses

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of POCD 7days after surgery | The seventh day after surgery

SECONDARY OUTCOMES:
Incidence of POCD 1 month after operation | One month after surgery
Incidence of POD 7 days after surgery | One day after surgery to the seventh day after surgery
  Use the CAM scale to assess whether a patient has postoperative delirium

CONTACTS AND LOCATIONS:
Overall Officials: su diansan, Study Chair — RenJi Hospital
Locations (3):
- China (3):
  - Renji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - Jin Cheng people's hospital, Jincheng, Shanxi

REFERENCES:
- [Derived] Zhang X, Chen Y, Tang Y, Zhang Y, Zhang X, Su D. Efficiency of probiotics in elderly patients undergoing orthopedic surgery for postoperative cognitive dysfunction: a study protocol for a multicenter, randomized controlled trial. Trials. 2023 Feb 25;24(1):146. doi: 10.1186/s13063-023-07167-6. PMID 36841790